CLINICAL TRIAL: NCT05180968
Title: Dialysis Symptom Control-Pruritus Outcome Trial: A Randomized Blinded Placebo Controlled Crossover Trial
Brief Title: DIalysis Symptom COntrol-Pruritus Outcome Trial
Acronym: DISCO-POT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Principal Investigator, David Collister, Adjunct Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2021:096
Record Dates: First submitted 2021-11-24; First posted 2022-01-06 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: End Stage Renal Disease; Pruritus
Keywords: Uremic; Pruritis; Itch; End Stage Renal Disease; Dialysis; Nabilone
MeSH Terms: conditions — Kidney Failure, Chronic; Pruritus | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nabilone 0.5mg (Experimental): Subjects will receive nabilone 0.5 mg orally at night for 1 week increased to nabilone 0.5mg orally twice a day for 3 weeks (over-encapsulated). Drug will be dispensed from a central site to other sites and pharmacy personnel will dispense the study medications directly to research personnel or participants. Drug dispensation will coincide with study visits at randomization and crossover and will allow research personnel to reinforced adherence. The study oral medications may be taken at any time of day with food or water, but we will request that participants take it at the same time each day, preferably at night when uremic pruritus symptoms are usually at the worst. If participants have any side effects or intolerability to study drugs, they may decrease the frequency of nabilone or placebo to 1 capsule by mouth once daily, preferably taken at night.
  Interventions: Drug: Nabilone 0.5 MG Oral Capsule
- Oral placebo (Placebo Comparator): Subjects will receive placebo 1 capsule orally at night for 1 week increased to placebo 2 capsules twice a day for 3 weeks (over-encapsulated). Drug will be dispensed from a central site to other sites and pharmacy personnel will dispense the study medications directly to research personnel or participants. Drug dispensation will coincide with study visits at randomization and crossover and will allow research personnel to reinforced adherence. The study oral medications may be taken at any time of day with food or water, but we will request that participants take it at the same time each day, preferably at night when uremic pruritus symptoms are usually at the worst. If participants have any side effects or intolerability to study drugs, they may decrease the frequency of nabilone or placebo to 1 capsule by mouth once daily, preferably taken at night.
  Interventions: Drug: Placebo Nabilone

INTERVENTIONS:
Drug: Nabilone 0.5 MG Oral Capsule — This intervention will consist of subjects receiving nabilone 0.5 mg orally at night for 1 week increased to nabilone 0.5mg orally twice a day for 3 weeks. Duration of the intervention will be 4 weeks.
  Other Names: TEVA-Nabilone
  Arms: Nabilone 0.5mg
Drug: Placebo Nabilone — This intervention will consist of subjects receiving placebo 1 capsule orally at night for 1 week increased to placebo 2 capsules twice a day for 3 weeks. Duration of the intervention will be 4 weeks.
  Other Names: TEVA-Nabilone Placebo
  Arms: Oral placebo

SUMMARY:
The purpose of this study is to test whether or not a medication called nabilone, which is a synthetic (non-natural) medication derived from cannabis, compared to placebo improves symptoms of itch in hemodialysis as measured by visual analog scales.

DETAILED DESCRIPTION:
Several different types of medications are effective in treating uremic pruritus, but even with effective treatments, residual symptoms are common and some medications are not well tolerated. Standard of care treatments include emollients which are lotions that keep the skin hydrated and a variety of pills that target the itch pathways implicated in the disease.

The objective of the study is to determine the proportion of patients with kidney failure for whom oral nabilone provides important benefit in reducing uremic pruritis without important adverse effects. The hypothesis is that there is a substantial proportion of patients in whom oral nabilone are safe and effective beyond placebo effects.

Nabilone is currently used to treat conditions other that uremic pruritus including chronic nerve pain as well as nausea and vomiting due to chemotherapy. It has never been studied in the setting of kidney disease.

DISCO-POT is a blinded, placebo-controlled crossover trial in which participants will be followed for 11 weeks including two 4 week treatment crossover periods with a 2 week washout period in between them and an end of study visit after 1 week off study drugs.

Patients that are eligible will be randomly assigned to a crossover treatment sequence of two treatments:

1. nabilone 0.5 mg orally at night for 1 week increased to nabilone 0.5mg orally twice a day for 3 weeks (over-encapsulated)
2. placebo 1 capsule orally at night for 1 week increased to placebo 2 capsules twice a day for 3 weeks (over-encapsulated)

ELIGIBILITY:
Inclusion Criteria:

1. Age>25 years
2. In-center or home hemodialysis at least two times weekly or peritoneal dialysis at least once daily for >90 days
3. Generalized uremic pruritus with a mean worst VAS>40mm over the previous week (with at least 5/7 patient diary days completed)
4. ALT less or equal to 3x upper limit of normal and bilirubin less than or equal to 2x upper limit of normal in the last 90 days
5. Able to provide informed consent and complete patient reported outcome measurements without a language barrier or cognitive impairment

Exclusion Criteria:

1. Etiology of pruritus (in the opinion of the treating physician) thought to be secondary to primary dermatologic condition, liver disease, hematologic malignancy or allergy
2. Use of recreational or medical cannabis in the last 4 weeks (THC, CBD, nabilone, Sativex, Epidiolex)
3. Women of childbearing potential as assessed by their clinician regardless of abstinence from sex or the use of contraception
4. Planned kidney transplantation, travel or relocation in the next 3 months
5. Unstable psychiatric illness (the presence of a lifetime diagnosis of a psychotic disorder, bipolar disorder, substance use disorder or current suicidal ideation)
6. Symptomatic hypotension in the last 2 weeks defined as a systolic blood pressure (SBP) less than 90mmHg during or in between dialysis requiring an intervention (i.e. administration of crystalloid or colloid, termination of dialysis, change in pharmacologic therapy such as withdrawal of anti-hypertensive therapy or initiation/titration of midodrine, increase in dry weight)
7. History of hypersensitivity to any cannabinoid
8. Presence of any clinically significant or unstable medical conditions, including cardiovascular, liver, pulmonary disease

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in worst uremic pruritis severity rating between treatment arms relative to MID | Measured at study baseline and weeks 1,2,3,4,5,6,7,8,9,10
  Measured using Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Number of participants with safety outcomes including adverse events related to study drug | Measured at study baseline and weeks 1,2,3,4,5,6,7,8,9,10,11
  serious adverse events, adverse events leading to drug discontinuation, hospitalization or emergency room visit for altered level of consciousness, fall, fracture, death, symptomatic hypotension requiring an intervention
Change in uremic pruritis severity | Measured at study baseline and weeks 1,2,3,4,5,6,7,8,9,10
  Measured as change from baseline in mean Visual Analogue Scale (VAS)
Change in uremic pruritis severity | Measured at study baseline and weeks 1,2,3,4,5,6,7,8,9,10
  Measured as change from baseline in mean Verbal Rating Scale (VRS)
Change in health-related quality of life | Measured at study baseline and weeks 3 and 4 of each crossover
  Measured using the Dermatology Quality of Life Index (DLQI)
Change in health-related quality of life | Measured at study baseline and weeks 3 and 4 of each crossover
  Measured using the EQ-5D 5 Level (EQ-5D-5L)
Change in health-related quality of life | Measured at study baseline and weeks 3 and 4 of each crossover
  Measured using the Patient Global Impression (PGI)
Effect of nabilone on sleep quality | Measured at study baseline and weeks 3 and 4 of each crossover
  Measured using the Pittsburgh Sleep Quality Index (PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: David Collister, MD, PhD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Seven Oaks General Hospital, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No